CLINICAL TRIAL: NCT01624142
Title: A Multicenter, Open-label Study to Assess the Long-term Safety, Tolerability, and Efficacy of Evolocumab (AMG145) on LDL-C in Subjects With Severe Familial Hypercholesterolemia
Brief Title: Trial Assessing Long Term USe of PCSK9 Inhibition in Subjects With Genetic LDL Disorders
Acronym: TAUSSIG
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20110271; 2011-005400-15 (EudraCT Number)
Record Dates: First submitted 2012-06-05; First posted 2012-06-20 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Severe Familial Hypercholesterolemia
Keywords: Hypercholesterolemia; Elevated Cholesterol; High Cholesterol; Homozygous Familial Hypercholesterolemia; PCSK9 mutations; Severe Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hypercholesterolemia; Homozygous Familial Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Evolocumab (Experimental): Participants received 420 mg evolocumab every month (participants not on lipid apheresis) or every 2 weeks (participants on lipid apheresis) for up to 5 years. Participants could switch dosing regimens at week 12 or 24 based on LDL-C and serum unbound proprotein convertase subtilisin/kexin type 9 (PCSK9) levels.
  Interventions: Biological: Evolocumab

INTERVENTIONS:
Biological: Evolocumab — Evolocumab was administered by subcutaneous injection either once a month (QM) or once every two weeks (Q2W).
  Other Names: AMG 145; Repatha

SUMMARY:
A study to assess the long term safety and tolerability of evolocumab (AMG 145) in adolescents and adults with severe familial hypercholesterolemia.

DETAILED DESCRIPTION:
This phase 2/3 open-label extension study was designed to characterize the safety and tolerability of long-term administration of evolocumab to adults and adolescents with severe FH (HoFH or non-HoFH severe FH). Participants not on lipid apheresis at enrollment or within the prior 8 weeks initiated treatment with evolocumab 420 mg once monthly (QM). Participants on lipid apheresis at enrollment initiated treatment with evolocumab 420 mg once every 2 weeks (Q2W). Dose frequency changes (420 mg QM vs 420 mg Q2W) were permitted at week 12, 24, or other visits with Sponsor approval. Participants with < 5% LDL-C reduction from baseline and serum unbound proprotein convertase subtilisin/kexin type 9 (PCSK9) < 100 ng/mL could discontinue evolocumab. If serum unbound PCSK9 was ≥ 100 ng/mL with QM dosing, the participant could switch to evolocumab 420 mg Q2W treatment. Participants on apheresis with ≥ 5% LDL-C reduction from baseline and serum unbound PCSK9 < 100 ng/mL with Q2W treatment could switch to QM dosing.

Participants were to continue to receive open-label evolocumab for up to 5 years or until evolocumab became commercially available in the relevant patient population, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

- Participated in Study 20110233 (NCT01588496) or another qualifying evolocumab parent protocol and have a diagnosis of familial hypercholesterolemia.

OR

* Have a diagnosis of familial hypercholesterolemia AND
* Males and females ≥ 12 to ≤ 80 years of age
* Stable low-fat diet and lipid-lowering therapies for at least 4 weeks
* Low-density lipoprotein cholesterol (LDL-C) >= 130 mg/dl (3.4 mmol/L) for subjects without diagnosed coronary heart disease (CHD)/CHD risk equivalent OR LDL-C >= 100 mg/dl (2.6 mmol/L) for subjects with diagnosed CHD or CHD risk equivalent OR apheresis patients have no LDL-C entry requirement
* Fasting triglycerides ≤ 400 mg/dL(4.5 mmol/L)
* Body weight of > 40 kg or greater at screening for subjects less than 18 years of age

Exclusion Criteria:

* New York Heart Failure Association (NYHA) class III or IV or last known left ventricular ejection fraction < 30%
* Myocardial infarction, unstable angina, percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or stroke within 3 months of screening
* Planned cardiac surgery or revascularization
* Uncontrolled cardiac arrhythmia
* Uncontrolled hypertension

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (41):
- United States (4):
  - Research Site, Los Angeles, California
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Nashville, Tennessee
- Australia (2):
  - Research Site, Hobart, Tasmania
  - Research Site, Perth, Western Australia
- Belgium (2):
  - Research Site, Brussels
  - Research Site, La Louvière
- Brazil (2):
  - Research Site, São Paulo, São Paulo
  - Research Site, São Paulo
- Canada (4):
  - Research Site, London, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Czechia (5):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
  - Research Site, Uherské Hradiště
- France (2):
  - Research Site, Dijon
  - Research Site, Paris
- Research Site, Athens, Greece
- Research Site, New Territories, Hong Kong
- Research Site, Ramat Gan, Israel
- Italy (3):
  - Research Site, Cinisello Balsamo (MI)
  - Research Site, Napoli
  - Research Site, Pisa
- Japan (2):
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Suita, Osaka
- Research Site, Beirut, Lebanon
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Rotterdam
- Research Site, Christchurch, New Zealand
- South Africa (2):
  - Research Site, Johannesburg, Gauteng
  - Research Site, Observatory, Western Cape
- Spain (5):
  - Research Site, Córdoba, Andalusia
  - Research Site, Barcelona, Catalonia
  - Research Site, A Coruña, Galicia
  - Research Site, Lugo, Galicia
  - Research Site, Madrid
- Research Site, Manchester, United Kingdom

REFERENCES:
- [Background] Raal FJ, Hovingh GK, Blom D, Santos RD, Harada-Shiba M, Bruckert E, Couture P, Soran H, Watts GF, Kurtz C, Honarpour N, Tang L, Kasichayanula S, Wasserman SM, Stein EA. Long-term treatment with evolocumab added to conventional drug therapy, with or without apheresis, in patients with homozygous familial hypercholesterolaemia: an interim subset analysis of the open-label TAUSSIG study. Lancet Diabetes Endocrinol. 2017 Apr;5(4):280-290. doi: 10.1016/S2213-8587(17)30044-X. Epub 2017 Feb 16. PMID 28215937
- [Background] Kasichayanula S, Grover A, Emery MG, Gibbs MA, Somaratne R, Wasserman SM, Gibbs JP. Clinical Pharmacokinetics and Pharmacodynamics of Evolocumab, a PCSK9 Inhibitor. Clin Pharmacokinet. 2018 Jul;57(7):769-779. doi: 10.1007/s40262-017-0620-7. PMID 29353350
- [Background] Santos RD, Stein EA, Hovingh GK, Blom DJ, Soran H, Watts GF, Lopez JAG, Bray S, Kurtz CE, Hamer AW, Raal FJ. Long-Term Evolocumab in Patients With Familial Hypercholesterolemia. J Am Coll Cardiol. 2020 Feb 18;75(6):565-574. doi: 10.1016/j.jacc.2019.12.020. PMID 32057369
- [Background] Raal FJ, Hegele RA, Ruzza A, Lopez JAG, Bhatia AK, Wu J, Wang H, Gaudet D, Wiegman A, Wang J, Santos RD. Evolocumab Treatment in Pediatric Patients With Homozygous Familial Hypercholesterolemia: Pooled Data From Three Open-Label Studies. Arterioscler Thromb Vasc Biol. 2024 May;44(5):1156-1164. doi: 10.1161/ATVBAHA.123.320268. Epub 2024 Mar 28. PMID 38545781
- [Derived] Schmidt AF, Carter JL, Pearce LS, Wilkins JT, Overington JP, Hingorani AD, Casas JP. PCSK9 monoclonal antibodies for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD011748. doi: 10.1002/14651858.CD011748.pub3. PMID 33078867
- [Derived] Stein EA, Honarpour N, Wasserman SM, Xu F, Scott R, Raal FJ. Effect of the proprotein convertase subtilisin/kexin 9 monoclonal antibody, AMG 145, in homozygous familial hypercholesterolemia. Circulation. 2013 Nov 5;128(19):2113-20. doi: 10.1161/CIRCULATIONAHA.113.004678. Epub 2013 Sep 6. PMID 24014831
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 43 centers in Canada, South Africa, Czech Republic, Netherlands, USA, France, Spain, Italy, Belgium, Australia, New Zealand, United Kingdom, Japan, Israel, Greece, Lebanon, Brazil, and Hong Kong between 01 June 2012 and 19 March 2015.
Pre-assignment Details: A total of 246 participants enrolled directly in Study 20110271 and 54 participants rolled over from Study 20110233 (NCT01588496).
  Results are reported separately for participants with homozygous familial hypercholesterolemia (HoFH) and non-HoFH severe familial hypercholesterolemia (FH) (ie, all those not meeting the protocol criteria for HoFH).
Groups:
- HoFH: Participants with homozygous familial hypercholesterolemia (HoFH) received 420 mg evolocumab every month (participants not on lipid apheresis) or every 2 weeks (participants on lipid apheresis) for up to 5 years. Participants could switch dosing regimens at week 12 or 24 based on LDL-C and serum unbound proprotein convertase subtilisin/kexin type 9 (PCSK9) levels.
- Severe FH: Participants with severe (non-HoFH) familial hypercholesterolemia (FH) received 420 mg evolocumab every month (participants not on lipid apheresis) or every 2 weeks (participants on lipid apheresis) for up to 5 years. Participants could switch dosing regimens at week 12 or 24 based on LDL-C and serum unbound PCSK9 levels.
Period: Overall Study
Arm/Group | HoFH | Severe FH
Started | 106 | 194
Completed | 74 | 178
Not Completed | 32 | 16
Not completed — Withdrawal by Subject | 14 | 4
Not completed — Death | 3 | 6
Not completed — Study Closure | 12 | 6
Not completed — Lost to Follow-up | 2 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants. Baseline data for parent study rollover participants are defined at the parent study baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | HoFH | Severe FH | Total
Number analyzed (Participants) | 106 | 194 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 0 | 14
  Between 18 and 65 years | 88 | 152 | 240
  >=65 years | 4 | 42 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (14.4) | 54.7 (11.9) | 47.5 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 78 | 132
  Male | 52 | 116 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 22 | 27
  Not Hispanic or Latino | 101 | 172 | 273
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 13 | 3 | 16
  Black or African American | 0 | 6 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 85 | 179 | 264
  Other | 7 | 4 | 11
  Mixed Race | 0 | 2 | 2
Low-density Lipoprotein Cholesterol (LDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 329.0 (136.7) | 192.7 (64.6) | 240.9 (116.3)
Non-high-density Lipoprotein Cholesterol (non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 350.5 (138.4) | 222.1 (68.3) | 267.5 (116.3)
Lipoprotein (a) Concentration [Mean (Standard Deviation); unit: nmol/L] | 104.7 (100.6) | 127.1 (142.8) | 119.2 (129.7)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] | 200.7 (69.9) | 139.2 (35.6) | 160.9 (58.3)
Total Cholesterol/HDL-C Ratio [Mean (Standard Deviation); unit: ratio] | 11.473 (6.312) | 6.055 (2.397) | 7.970 (4.943)
Apolipoprotein B/Apoliprotein A1 Ratio [Mean (Standard Deviation); unit: ratio] | 1.984 (0.950) | 1.023 (0.355) | 1.362 (0.781)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The severity of each adverse event (AE) was graded according to the National Cancer Institute Common Terminology Criteria for AEs (NCI-CTCAE) grading scale, where grade 1 = mild AE, grade 2 = moderate AE, grade 3 = severe AE, grade 4 = life-threatening AE and grade 5 = death due to AE.
Time Frame: From first dose of study drug in Study 20110271 up to 30 days after the last dose or until the end of study date, whichever was earlier; median duration of treatment was 48.7 months.
Population: All participants who received at least one dose of evolocumab in Study 20110271
Measure: Count of Participants; unit: Participants
Arm/Group | HoFH | Severe FH
Number analyzed (Participants) | 106 | 194
Participants
  All adverse events (AEs) | 94 | 174
  Adverse events ≥ grade 2 | 76 | 143
  Adverse events ≥ grade 3 | 38 | 68
  Adverse events ≥ grade 4 | 4 | 14
  Serious adverse events (SAEs) | 29 | 57
  AEs Leading to discontinuation of evolocumab | 3 | 8
  Fatal adverse events | 2 | 5
  Device-related adverse events | 6 | 18

2. Secondary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C)
Time Frame: Baseline and weeks 4, 6, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, and 216
Population: Participants who received at least 1 dose of evolocumab in Study 20110271 and with available data at each time point.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | HoFH | Severe FH
Number analyzed (Participants) | 106 | 194
percent change
  Week 4: number analyzed (Participants) | 87 | 183
  Week 4 | -20.42 [-38.25 to -8.28] | -54.95 [-66.67 to -44.55]
  Week 6: number analyzed (Participants) | 83 | 166
  Week 6 | -18.32 [-36.09 to -4.16] | -67.57 [-79.54 to -53.93]
  Week 8: number analyzed (Participants) | 94 | 187
  Week 8 | -20.28 [-37.81 to -8.44] | -55.03 [-68.58 to -42.07]
  Week 12: number analyzed (Participants) | 104 | 191
  Week 12 | -18.26 [-36.06 to -7.76] | -57.11 [-68.00 to -42.80]
  Week 16: number analyzed (Participants) | 102 | 188
  Week 16 | -23.15 [-39.23 to -7.87] | -57.53 [-67.99 to -44.95]
  Week 20: number analyzed (Participants) | 101 | 185
  Week 20 | -25.37 [-45.99 to -8.96] | -57.26 [-67.48 to -44.68]
  Week 24: number analyzed (Participants) | 99 | 191
  Week 24 | -21.84 [-41.39 to -8.11] | -57.10 [-67.05 to -43.70]
  Week 36: number analyzed (Participants) | 94 | 187
  Week 36 | -26.79 [-46.44 to -8.28] | -56.08 [-68.70 to -44.47]
  Week 48: number analyzed (Participants) | 93 | 187
  Week 48 | -25.50 [-44.79 to -4.43] | -59.67 [-69.14 to -47.88]
  Week 60: number analyzed (Participants) | 88 | 186
  Week 60 | -27.26 [-44.58 to -4.28] | -57.13 [-68.42 to -42.65]
  Week 72: number analyzed (Participants) | 85 | 184
  Week 72 | -27.11 [-51.06 to -12.03] | -55.73 [-70.52 to -42.76]
  Week 84: number analyzed (Participants) | 82 | 180
  Week 84 | -27.96 [-50.29 to -7.96] | -56.02 [-68.49 to -42.18]
  Week 96: number analyzed (Participants) | 82 | 180
  Week 96 | -22.47 [-46.53 to -8.12] | -57.10 [-69.53 to -41.66]
  Week 108: number analyzed (Participants) | 82 | 181
  Week 108 | -26.15 [-44.58 to -5.62] | -60.57 [-69.47 to -43.15]
  Week 120: number analyzed (Participants) | 82 | 184
  Week 120 | -26.66 [-43.43 to -7.42] | -56.76 [-69.48 to -41.70]
  Week 132: number analyzed (Participants) | 81 | 177
  Week 132 | -28.25 [-48.23 to -9.42] | -55.25 [-68.17 to -39.89]
  Week 144: number analyzed (Participants) | 79 | 180
  Week 144 | -28.33 [-49.27 to -10.33] | -56.48 [-69.26 to -40.69]
  Week 156: number analyzed (Participants) | 80 | 181
  Week 156 | -23.65 [-47.66 to -11.05] | -55.38 [-69.48 to -41.03]
  Week 168: number analyzed (Participants) | 76 | 171
  Week 168 | -29.52 [-51.35 to -4.41] | -54.77 [-67.16 to -36.42]
  Week 180: number analyzed (Participants) | 74 | 166
  Week 180 | -25.66 [-53.71 to -9.87] | -54.08 [-71.53 to -37.55]
  Week 192: number analyzed (Participants) | 74 | 147
  Week 192 | -30.12 [-53.23 to -11.81] | -52.19 [-66.79 to -33.99]
  Week 204: number analyzed (Participants) | 75 | 129
  Week 204 | -29.62 [-47.43 to -6.11] | -59.59 [-70.50 to -39.06]
  Week 216: number analyzed (Participants) | 68 | 96
  Week 216 | -32.22 [-46.65 to -8.97] | -50.62 [-67.73 to -32.31]

3. Secondary Outcome: Percent Change From Baseline in Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Time Frame: as for outcome 2
Population: Participants who received at least 1 dose of evolocumab in Study 20110271 and with available data at each time point.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | HoFH | Severe FH
Number analyzed (Participants) | 106 | 194
percent change
  Week 4: number analyzed (Participants) | 88 | 183
  Week 4 | -19.62 [-35.54 to -7.84] | -50.00 [-59.92 to -39.88]
  Week 6: number analyzed (Participants) | 85 | 168
  Week 6 | -18.17 [-33.88 to -4.29] | -59.76 [-70.50 to -49.23]
  Week 8: number analyzed (Participants) | 94 | 188
  Week 8 | -20.29 [-35.94 to -9.28] | -50.61 [-58.49 to -37.91]
  Week 12: number analyzed (Participants) | 105 | 192
  Week 12 | -17.05 [-32.03 to -6.99] | -50.25 [-61.49 to -38.63]
  Week 16: number analyzed (Participants) | 102 | 188
  Week 16 | -21.73 [-37.81 to -7.88] | -51.31 [-59.76 to -40.40]
  Week 20: number analyzed (Participants) | 101 | 188
  Week 20 | -24.09 [-43.06 to -7.76] | -50.76 [-59.44 to -38.67]
  Week 24: number analyzed (Participants) | 100 | 192
  Week 24 | -21.88 [-38.81 to -9.54] | -51.12 [-60.67 to -38.52]
  Week 36: number analyzed (Participants) | 95 | 190
  Week 36 | -22.43 [-44.08 to -6.22] | -49.65 [-61.00 to -38.26]
  Week 48: number analyzed (Participants) | 94 | 190
  Week 48 | -24.08 [-43.47 to -3.98] | -51.12 [-61.58 to -42.11]
  Week 60: number analyzed (Participants) | 89 | 189
  Week 60 | -24.81 [-42.96 to -2.67] | -49.73 [-61.61 to -38.00]
  Week 72: number analyzed (Participants) | 85 | 188
  Week 72 | -25.88 [-48.21 to -9.47] | -48.94 [-61.14 to -36.08]
  Week 84: number analyzed (Participants) | 83 | 184
  Week 84 | -21.00 [-42.68 to -7.45] | -49.50 [-62.07 to -35.14]
  Week 96: number analyzed (Participants) | 83 | 184
  Week 96 | -21.10 [-42.84 to -7.85] | -49.53 [-63.80 to -36.86]
  Week 108: number analyzed (Participants) | 83 | 186
  Week 108 | -24.17 [-43.01 to -5.69] | -52.86 [-61.20 to -38.11]
  Week 120: number analyzed (Participants) | 82 | 185
  Week 120 | -23.21 [-40.37 to -6.23] | -49.45 [-60.48 to -35.91]
  Week 132: number analyzed (Participants) | 82 | 182
  Week 132 | -26.39 [-40.28 to -7.19] | -49.49 [-60.95 to -33.66]
  Week 144: number analyzed (Participants) | 81 | 183
  Week 144 | -25.38 [-45.55 to -8.08] | -49.81 [-61.69 to -33.88]
  Week 156: number analyzed (Participants) | 80 | 184
  Week 156 | -22.35 [-45.47 to -10.50] | -50.15 [-60.81 to -36.11]
  Week 168: number analyzed (Participants) | 76 | 176
  Week 168 | -27.97 [-48.82 to -4.36] | -47.93 [-60.71 to -31.01]
  Week 180: number analyzed (Participants) | 74 | 167
  Week 180 | -26.32 [-49.82 to -8.62] | -48.43 [-62.22 to -33.06]
  Week 192: number analyzed (Participants) | 75 | 151
  Week 192 | -27.61 [-49.49 to -9.29] | -44.50 [-57.71 to -29.77]
  Week 204: number analyzed (Participants) | 75 | 131
  Week 204 | -27.22 [-45.14 to -5.73] | -50.84 [-64.12 to -36.03]
  Week 216: number analyzed (Participants) | 68 | 98
  Week 216 | -31.40 [-42.75 to -9.67] | -45.30 [-61.45 to -26.32]

4. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a)
Time Frame: as for outcome 2
Population: Participants who received at least 1 dose of evolocumab in Study 20110271 and with available data at each time point.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | HoFH | Severe FH
Number analyzed (Participants) | 106 | 194
percent change
  Week 4: number analyzed (Participants) | 87 | 183
  Week 4 | -11.11 [-27.50 to 0.0] | -20.49 [-39.84 to -11.61]
  Week 6: number analyzed (Participants) | 85 | 169
  Week 6 | -8.97 [-24.21 to 3.76] | -24.42 [-45.95 to -9.38]
  Week 8: number analyzed (Participants) | 94 | 188
  Week 8 | -9.95 [-25.00 to 3.23] | -21.51 [-39.84 to -9.09]
  Week 12: number analyzed (Participants) | 105 | 192
  Week 12 | -7.69 [-21.64 to 6.83] | -24.40 [-40.28 to -9.09]
  Week 16: number analyzed (Participants) | 103 | 188
  Week 16 | -8.93 [-25.00 to 4.76] | -23.08 [-38.88 to -7.62]
  Week 20: number analyzed (Participants) | 100 | 188
  Week 20 | -13.52 [-29.36 to 0.00] | -22.21 [-39.34 to -5.98]
  Week 24: number analyzed (Participants) | 100 | 192
  Week 24 | -10.46 [-23.75 to 1.00] | -25.99 [-41.81 to -9.09]
  Week 36: number analyzed (Participants) | 95 | 190
  Week 36 | -15.14 [-28.18 to 0.00] | -24.26 [-41.30 to -7.85]
  Week 48: number analyzed (Participants) | 94 | 189
  Week 48 | -13.17 [-30.51 to 0.00] | -26.32 [-41.94 to -10.49]
  Week 60: number analyzed (Participants) | 90 | 189
  Week 60 | -13.04 [-35.00 to 2.86] | -24.05 [-41.97 to -7.63]
  Week 72: number analyzed (Participants) | 86 | 188
  Week 72 | -17.43 [-37.19 to 5.88] | -24.23 [-43.96 to -6.81]
  Week 84: number analyzed (Participants) | 84 | 184
  Week 84 | -14.12 [-36.73 to 0.63] | -24.12 [-44.05 to -8.02]
  Week 96: number analyzed (Participants) | 83 | 184
  Week 96 | -17.24 [-33.33 to 0.49] | -31.28 [-47.33 to -13.34]
  Week 108: number analyzed (Participants) | 83 | 186
  Week 108 | -21.43 [-42.50 to 0.00] | -32.44 [-48.65 to -12.69]
  Week 120: number analyzed (Participants) | 82 | 186
  Week 120 | -20.16 [-33.25 to 0.00] | -31.22 [-45.00 to -11.40]
  Week 132: number analyzed (Participants) | 82 | 182
  Week 132 | -19.15 [-37.68 to 0.00] | -29.32 [-49.82 to -12.29]
  Week 144: number analyzed (Participants) | 81 | 183
  Week 144 | -23.64 [-47.06 to 0.00] | -30.36 [-48.17 to -11.92]
  Week 156: number analyzed (Participants) | 80 | 184
  Week 156 | -18.40 [-42.14 to -2.33] | -28.10 [-47.35 to -9.09]
  Week 168: number analyzed (Participants) | 76 | 176
  Week 168 | -22.94 [-41.01 to -0.49] | -23.96 [-45.64 to -9.09]
  Week 180: number analyzed (Participants) | 74 | 168
  Week 180 | -17.29 [-43.83 to 0.00] | -26.23 [-46.01 to -8.83]
  Week 192: number analyzed (Participants) | 75 | 151
  Week 192 | -22.78 [-44.44 to 0.00] | -20.00 [-37.75 to -2.44]
  Week 204: number analyzed (Participants) | 75 | 131
  Week 204 | -16.33 [-38.46 to 3.95] | -14.29 [-34.38 to 10.00]
  Week 216: number analyzed (Participants) | 68 | 98
  Week 216 | -14.06 [-36.07 to 4.08] | -0.67 [-23.64 to 23.81]

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B
Time Frame: as for outcome 2
Population: Participants who received at least 1 dose of evolocumab in Study 20110271 and with available data at each time point.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | HoFH | Severe FH
Number analyzed (Participants) | 106 | 194
percent change
  Week 4: number analyzed (Participants) | 88 | 183
  Week 4 | -16.91 [-31.67 to -6.81] | -43.84 [-54.59 to -34.40]
  Week 6: number analyzed (Participants) | 85 | 169
  Week 6 | -16.25 [-27.82 to -1.96] | -56.70 [-67.23 to -46.11]
  Week 8: number analyzed (Participants) | 94 | 188
  Week 8 | -17.57 [-32.00 to -6.24] | -43.95 [-55.69 to -31.55]
  Week 12: number analyzed (Participants) | 105 | 192
  Week 12 | -13.11 [-26.87 to -3.49] | -45.78 [-55.16 to -32.65]
  Week 16: number analyzed (Participants) | 102 | 188
  Week 16 | -18.65 [-34.77 to -8.35] | -45.72 [-55.23 to -35.39]
  Week 20: number analyzed (Participants) | 101 | 188
  Week 20 | -22.60 [-39.05 to -5.03] | -45.16 [-53.93 to -33.18]
  Week 24: number analyzed (Participants) | 100 | 192
  Week 24 | -20.09 [-33.04 to -3.97] | -44.87 [-55.32 to -31.01]
  Week 36: number analyzed (Participants) | 95 | 190
  Week 36 | -16.48 [-36.43 to -2.56] | -43.33 [-55.12 to -29.10]
  Week 48: number analyzed (Participants) | 94 | 190
  Week 48 | -15.90 [-33.60 to -4.15] | -45.38 [-55.40 to -33.93]
  Week 60: number analyzed (Participants) | 90 | 189
  Week 60 | -15.99 [-38.12 to -0.27] | -44.81 [-56.07 to -31.33]
  Week 72: number analyzed (Participants) | 86 | 188
  Week 72 | -20.70 [-42.02 to -3.17] | -44.07 [-55.61 to -32.72]
  Week 84: number analyzed (Participants) | 84 | 184
  Week 84 | -19.52 [-35.66 to -0.09] | -43.87 [-55.50 to -32.13]
  Week 96: number analyzed (Participants) | 83 | 184
  Week 96 | -15.07 [-36.34 to -3.67] | -42.31 [-57.65 to -29.89]
  Week 108: number analyzed (Participants) | 83 | 186
  Week 108 | -19.45 [-36.07 to 5.03] | -46.30 [-55.41 to -32.21]
  Week 120: number analyzed (Participants) | 82 | 185
  Week 120 | -21.58 [-33.33 to -1.57] | -44.33 [-54.68 to -30.00]
  Week 132: number analyzed (Participants) | 82 | 181
  Week 132 | -22.44 [-35.70 to -3.75] | -43.48 [-54.90 to -28.22]
  Week 144: number analyzed (Participants) | 81 | 183
  Week 144 | -21.24 [-41.89 to -3.55] | -41.64 [-54.36 to -27.85]
  Week 156: number analyzed (Participants) | 80 | 184
  Week 156 | -18.30 [-36.66 to -5.63] | -44.04 [-55.16 to -29.73]
  Week 168: number analyzed (Participants) | 76 | 176
  Week 168 | -20.38 [-41.58 to -2.81] | -40.20 [-52.22 to -25.78]
  Week 180: number analyzed (Participants) | 74 | 168
  Week 180 | -19.51 [-39.73 to -3.02] | -41.58 [-54.70 to -24.57]
  Week 192: number analyzed (Participants) | 75 | 151
  Week 192 | -19.38 [-39.63 to -2.63] | -37.02 [-52.06 to -21.08]
  Week 204: number analyzed (Participants) | 75 | 131
  Week 204 | -21.64 [-36.15 to -5.48] | -43.19 [-56.81 to -28.81]
  Week 216: number analyzed (Participants) | 68 | 98
  Week 216 | -22.68 [-35.34 to -4.51] | -35.95 [-53.05 to -23.95]

6. Secondary Outcome: Percent Change From Baseline in Total Cholesterol/HDL-C Ratio
Time Frame: as for outcome 2
Population: Participants who received at least 1 dose of evolocumab in Study 20110271 and with available data at each time point.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | HoFH | Severe FH
Number analyzed (Participants) | 106 | 194
percent change
  Week 4: number analyzed (Participants) | 88 | 183
  Week 4 | -21.32 [-38.45 to -10.36] | -43.49 [-53.07 to -33.78]
  Week 6: number analyzed (Participants) | 85 | 168
  Week 6 | -23.25 [-35.54 to -7.14] | -52.38 [-60.97 to -42.29]
  Week 8: number analyzed (Participants) | 94 | 188
  Week 8 | -23.93 [-35.26 to -5.42] | -43.44 [-51.21 to -34.81]
  Week 12: number analyzed (Participants) | 105 | 192
  Week 12 | -21.20 [-34.98 to -9.31] | -44.75 [-53.20 to -35.12]
  Week 16: number analyzed (Participants) | 102 | 188
  Week 16 | -24.01 [-36.52 to -8.86] | -45.31 [-52.38 to -34.95]
  Week 20: number analyzed (Participants) | 101 | 188
  Week 20 | -24.69 [-36.39 to -4.29] | -43.07 [-51.89 to -33.54]
  Week 24: number analyzed (Participants) | 100 | 192
  Week 24 | -23.53 [-38.59 to -9.10] | -43.79 [-52.96 to -34.28]
  Week 36: number analyzed (Participants) | 95 | 190
  Week 36 | -27.16 [-42.86 to -9.12] | -42.69 [-53.01 to -30.99]
  Week 48: number analyzed (Participants) | 94 | 190
  Week 48 | -26.54 [-43.73 to -8.03] | -44.68 [-54.47 to -33.90]
  Week 60: number analyzed (Participants) | 89 | 189
  Week 60 | -22.80 [-45.57 to -5.13] | -43.82 [-54.01 to -32.46]
  Week 72: number analyzed (Participants) | 85 | 188
  Week 72 | -24.79 [-42.72 to -9.47] | -42.64 [-54.28 to -30.73]
  Week 84: number analyzed (Participants) | 83 | 184
  Week 84 | -22.62 [-41.45 to -6.24] | -43.16 [-53.15 to -27.42]
  Week 96: number analyzed (Participants) | 83 | 184
  Week 96 | -23.00 [-38.97 to -10.33] | -42.46 [-54.03 to -31.69]
  Week 108: number analyzed (Participants) | 83 | 186
  Week 108 | -25.03 [-41.12 to -4.98] | -43.68 [-53.91 to -32.90]
  Week 120: number analyzed (Participants) | 82 | 185
  Week 120 | -25.40 [-42.55 to -6.92] | -42.42 [-54.18 to -30.87]
  Week 132: number analyzed (Participants) | 82 | 182
  Week 132 | -25.66 [-41.29 to -5.10] | -42.14 [-53.54 to -30.15]
  Week 144: number analyzed (Participants) | 81 | 183
  Week 144 | -27.79 [-44.96 to -6.39] | -43.40 [-54.91 to -28.80]
  Week 156: number analyzed (Participants) | 80 | 184
  Week 156 | -25.52 [-45.62 to -9.87] | -43.85 [-53.49 to -29.86]
  Week 168: number analyzed (Participants) | 76 | 176
  Week 168 | -26.30 [-46.28 to -8.75] | -41.59 [-52.67 to -24.39]
  Week 180: number analyzed (Participants) | 74 | 167
  Week 180 | -29.53 [-47.74 to -7.54] | -40.13 [-54.50 to -28.99]
  Week 192: number analyzed (Participants) | 75 | 151
  Week 192 | -27.79 [-47.16 to -12.15] | -38.24 [-53.80 to -25.34]
  Week 204: number analyzed (Participants) | 75 | 131
  Week 204 | -27.32 [-42.19 to -7.20] | -43.13 [-57.50 to -31.50]
  Week 216: number analyzed (Participants) | 68 | 98
  Week 216 | -30.92 [-42.09 to -8.93] | -40.78 [-52.60 to -26.46]

7. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A1 Ratio
Time Frame: as for outcome 2
Population: Participants who received at least 1 dose of evolocumab in Study 20110271 and with available data at each time point.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | HoFH | Severe FH
Number analyzed (Participants) | 106 | 194
percent change
  Week 4: number analyzed (Participants) | 88 | 183
  Week 4 | -23.06 [-39.88 to -6.22] | -46.79 [-57.95 to -37.69]
  Week 6: number analyzed (Participants) | 85 | 169
  Week 6 | -21.38 [-36.90 to -10.11] | -59.77 [-68.35 to -48.98]
  Week 8: number analyzed (Participants) | 94 | 188
  Week 8 | -21.53 [-36.51 to -4.66] | -47.82 [-57.87 to -37.07]
  Week 12: number analyzed (Participants) | 105 | 192
  Week 12 | -16.67 [-30.72 to -4.37] | -48.63 [-59.21 to -38.16]
  Week 16: number analyzed (Participants) | 102 | 188
  Week 16 | -22.52 [-42.86 to -8.97] | -48.98 [-58.13 to -39.59]
  Week 20: number analyzed (Participants) | 101 | 188
  Week 20 | -25.41 [-41.87 to -12.43] | -49.12 [-57.11 to -38.09]
  Week 24: number analyzed (Participants) | 100 | 192
  Week 24 | -22.97 [-38.08 to -8.99] | -49.92 [-58.44 to -37.29]
  Week 36: number analyzed (Participants) | 95 | 190
  Week 36 | -26.86 [-41.04 to -7.69] | -49.02 [-58.10 to -35.67]
  Week 48: number analyzed (Participants) | 94 | 190
  Week 48 | -25.96 [-43.38 to -12.26] | -49.35 [-59.34 to -38.98]
  Week 60: number analyzed (Participants) | 90 | 189
  Week 60 | -24.31 [-44.46 to -6.67] | -48.57 [-59.11 to -35.94]
  Week 72: number analyzed (Participants) | 86 | 188
  Week 72 | -23.63 [-45.15 to -10.89] | -48.94 [-60.36 to -38.76]
  Week 84: number analyzed (Participants) | 84 | 184
  Week 84 | -24.09 [-43.12 to -4.16] | -49.47 [-59.73 to -34.54]
  Week 96: number analyzed (Participants) | 83 | 184
  Week 96 | -24.75 [-45.92 to -8.61] | -48.45 [-60.40 to -36.17]
  Week 108: number analyzed (Participants) | 83 | 186
  Week 108 | -26.03 [-41.27 to -4.78] | -50.18 [-60.18 to -37.84]
  Week 120: number analyzed (Participants) | 82 | 185
  Week 120 | -26.45 [-44.21 to -12.32] | -49.75 [-59.38 to -36.17]
  Week 132: number analyzed (Participants) | 82 | 181
  Week 132 | -24.26 [-47.15 to -7.81] | -48.54 [-58.39 to -32.01]
  Week 144: number analyzed (Participants) | 81 | 183
  Week 144 | -28.09 [-48.50 to -7.81] | -47.44 [-59.12 to -33.82]
  Week 156: number analyzed (Participants) | 80 | 184
  Week 156 | -27.21 [-46.95 to -12.25] | -49.10 [-59.29 to -35.31]
  Week 168: number analyzed (Participants) | 76 | 176
  Week 168 | -32.16 [-47.39 to -12.53] | -44.46 [-56.03 to -30.06]
  Week 180: number analyzed (Participants) | 74 | 168
  Week 180 | -28.70 [-48.45 to -9.71] | -45.13 [-58.67 to -30.84]
  Week 192: number analyzed (Participants) | 75 | 151
  Week 192 | -27.50 [-50.49 to -10.22] | -43.40 [-56.45 to -28.14]
  Week 204: number analyzed (Participants) | 75 | 131
  Week 204 | -28.04 [-46.84 to -12.13] | -49.71 [-60.22 to -35.16]
  Week 216: number analyzed (Participants) | 68 | 98
  Week 216 | -28.37 [-41.15 to -11.76] | -44.00 [-56.69 to -31.29]

8. Secondary Outcome: Percentage of Participants With a 15% or Greater Reduction in LDL-C
Time Frame: as for outcome 2
Population: Participants who received at least 1 dose of evolocumab in Study 20110271 and with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | HoFH | Severe FH
Number analyzed (Participants) | 106 | 194
percentage of participants
  Week 4: number analyzed (Participants) | 87 | 183
  Week 4 | 62.1 | 98.9
  Week 6: number analyzed (Participants) | 83 | 166
  Week 6 | 51.8 | 98.2
  Week 8: number analyzed (Participants) | 94 | 187
  Week 8 | 57.4 | 97.9
  Week 12: number analyzed (Participants) | 104 | 191
  Week 12 | 56.7 | 99.0
  Week 16: number analyzed (Participants) | 102 | 188
  Week 16 | 63.7 | 97.3
  Week 20: number analyzed (Participants) | 101 | 185
  Week 20 | 64.4 | 98.9
  Week 24: number analyzed (Participants) | 99 | 191
  Week 24 | 66.7 | 96.3
  Week 36: number analyzed (Participants) | 94 | 187
  Week 36 | 62.8 | 97.3
  Week 48: number analyzed (Participants) | 93 | 187
  Week 48 | 60.2 | 97.9
  Week 60: number analyzed (Participants) | 88 | 186
  Week 60 | 60.2 | 94.1
  Week 72: number analyzed (Participants) | 85 | 184
  Week 72 | 69.4 | 94.0
  Week 84: number analyzed (Participants) | 82 | 180
  Week 84 | 65.9 | 93.9
  Week 96: number analyzed (Participants) | 82 | 180
  Week 96 | 65.9 | 94.4
  Week 108: number analyzed (Participants) | 82 | 181
  Week 108 | 61.0 | 96.1
  Week 120: number analyzed (Participants) | 82 | 184
  Week 120 | 64.6 | 91.8
  Week 132: number analyzed (Participants) | 81 | 177
  Week 132 | 61.7 | 92.7
  Week 144: number analyzed (Participants) | 79 | 180
  Week 144 | 72.2 | 93.3
  Week 156: number analyzed (Participants) | 80 | 181
  Week 156 | 68.8 | 93.4
  Week 168: number analyzed (Participants) | 76 | 171
  Week 168 | 59.2 | 93.6
  Week 180: number analyzed (Participants) | 74 | 166
  Week 180 | 63.5 | 93.4
  Week 192: number analyzed (Participants) | 74 | 147
  Week 192 | 66.2 | 91.8
  Week 204: number analyzed (Participants) | 75 | 129
  Week 204 | 65.3 | 93.8
  Week 216: number analyzed (Participants) | 68 | 96
  Week 216 | 70.6 | 88.5

ADVERSE EVENTS:
Time Frame: Adverse events are reported from the first dose of study drug in Study 20110271 up to 30 days after the last dose or until the end of study date, whichever was earlier; median duration of treatment was 48.7 months. Deaths are reported from the first dose of study drug up to the end of study visit date.
Description: In some cases the time frame between last dose and end of study visit was more than 30 days. Two participants in included in the all-cause mortality table died more than 30 days after last dose of study drug.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Total: Participants received 420 mg evolocumab every month (participants not on lipid apheresis) or every 2 weeks (participants on lipid apheresis) for up to 5 years. Participants could switch dosing regimens at week 12 or 24 based on LDL-C and serum unbound PCSK9 levels.
Arm/Group | HoFH | Severe FH | Total
All-Cause Mortality (participants affected / at risk) | 3/106 | 6/194 | 9/300
Serious Adverse Events (participants affected / at risk) | 29/106 | 57/194 | 86/300
Other Adverse Events (participants affected / at risk) | 80/106 | 134/194 | 214/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HoFH (N=106) | Severe FH (N=194) | Total (N=300)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 2 | 4
Angina pectoris (Cardiac disorders) | 4 | 7 | 11
Angina unstable (Cardiac disorders) | 0 | 3 | 3
Aortic valve disease (Cardiac disorders) | 1 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 3 | 1 | 4
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 4 | 5
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1
Supravalvular aortic stenosis (Cardiac disorders) | 1 | 0 | 1
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Cataract (Eye disorders) | 1 | 1 | 2
Glaucoma (Eye disorders) | 0 | 1 | 1
Macular degeneration (Eye disorders) | 0 | 1 | 1
Macular hole (Eye disorders) | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Gingival cyst (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 1
Chest discomfort (General disorders) | 1 | 0 | 1
Chest pain (General disorders) | 1 | 5 | 6
Complication associated with device (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 3 | 4
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 2
Hepatic cyst (Hepatobiliary disorders) | 0 | 1 | 1
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1 | 2
Diverticulitis (Infections and infestations) | 0 | 2 | 2
Osteomyelitis chronic (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 3
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1
Cardiac stress test abnormal (Investigations) | 0 | 1 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 1 | 1
Troponin increased (Investigations) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Ovarian germ cell teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Dementia with Lewy bodies (Nervous system disorders) | 0 | 1 | 1
Embolic stroke (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 2
Renal infarct (Renal and urinary disorders) | 0 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Aortic stenosis (Vascular disorders) | 3 | 2 | 5
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HoFH (N=106) | Severe FH (N=194) | Total (N=300)
Abdominal pain (Gastrointestinal disorders) | 7 | 7 | 14
Diarrhoea (Gastrointestinal disorders) | 7 | 22 | 29
Chest pain (General disorders) | 4 | 15 | 19
Fatigue (General disorders) | 8 | 19 | 27
Influenza like illness (General disorders) | 2 | 10 | 12
Injection site bruising (General disorders) | 4 | 10 | 14
Injection site pain (General disorders) | 6 | 5 | 11
Oedema peripheral (General disorders) | 3 | 11 | 14
Bronchitis (Infections and infestations) | 4 | 16 | 20
Gastroenteritis (Infections and infestations) | 6 | 12 | 18
Influenza (Infections and infestations) | 17 | 21 | 38
Nasopharyngitis (Infections and infestations) | 17 | 36 | 53
Sinusitis (Infections and infestations) | 7 | 7 | 14
Upper respiratory tract infection (Infections and infestations) | 18 | 17 | 35
Urinary tract infection (Infections and infestations) | 8 | 12 | 20
Alanine aminotransferase increased (Investigations) | 6 | 3 | 9
Blood creatine phosphokinase increased (Investigations) | 6 | 4 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 23 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 17 | 26
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 15 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 24 | 30
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 11 | 15
Dizziness (Nervous system disorders) | 4 | 12 | 16
Headache (Nervous system disorders) | 17 | 16 | 33
Anxiety (Psychiatric disorders) | 10 | 0 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 14 | 19
Hypertension (Vascular disorders) | 9 | 15 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2015-12-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT01624142/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT01624142/SAP_001.pdf